CLINICAL TRIAL: NCT01967303
Title: Restless Legs Syndrome in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Ilana Schlesinger, Director, Movement Disorders Center, Rambam Health Care Campus
Other Study IDs: 3186
Record Dates: First submitted 2013-09-15; First posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Restless Legs Syndrome; Stroke; Transient Ischemic Attack
Keywords: Restless legs syndrome; Stroke; Transient ischemic attack; Cerebrovascular risk factors
MeSH Terms: conditions — Restless Legs Syndrome; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with stroke or transient ischemic attack: Interview regarding restless legs syndrome
- Subjects without stroke or transient ischemic attack: Interview regarding restless legs syndrome

SUMMARY:
Our study aimed to examine a possible association between Restless legs syndrome and cerebrovascular disease, by examining patients during hospitalization for acute stroke or transient ischemic attack, in a matched case-control design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Hospitalization for stroke or transient ischemic attack

Exclusion Criteria:

* 18 years old or younger
* No stroke or transient ischemic attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with stroke or transient ischemic attack.
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of Restless legs syndrome in patients with stroke or Transient ischemic attack vs. prevalence in controls. | At time of interview
  The frequency (prevalence) of restless leg syndrome (RLS) in patients who have suffered stroke or TIA will be compared to that of subjects who have not suffered stroke or TIA (controls). The two groups will be stratified with regard to age and gender. Statistical comparison will be made by univariate analyses and by multivariate logistic regression analyses (which will include cerebrovascular risk factors besides stroke or TIA).

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Schlesinger, Principal Investigator — Rambam Health Care Campus, Haifa, Israel